CLINICAL TRIAL: NCT02821130
Title: Effects of Orkambi on Exertional Dyspnea, Exercise Performance, and Ventilatory Responses in Adults With Cystic Fibrosis
Brief Title: Orkambi Exercise Study
Acronym: Orkambi
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Assistant Professor, University of British Columbia
Other Study IDs: H16-01164
Record Dates: First submitted 2016-06-06; First posted 2016-07-01 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Lung; Disease; Cystic Fibrosis
Keywords: Dyspnea; Exercise; Cystic Fibrosis
MeSH Terms: conditions — Lung Diseases; Cystic Fibrosis; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis Patients: Participants diagnosed with cystic fibrosis

SUMMARY:
Shortness of breath (dyspnea) during exercise is a major source of distress and is a commonly reported symptom in patients with cystic fibrosis (CF). A recent treatment option known as Orkambi, which combines the drugs lumacaftor and ivacaftor, may be used in patients with CF to help improve lung health. However, the effects of this combination therapy on dyspnea and exercise performance, a known predictor of survival in CF, are not clear. The investigators aim to understand the effects of Orkambi on these symptoms and to gain new insight into the potential health improvements in CF from using this treatment option.

DETAILED DESCRIPTION:
Advances in therapies and patient care have led to dramatic improvements in cystic fibrosis (CF) survival. Consequently, CF patients are living longer with varying degrees of lung function impairment. Dyspnea is a commonly reported symptom in CF that adversely impacts quality of life. Recently, lumacaftor/ivacaftor (Orkambi), a combination drug therapy, was approved by Health Canada for use in CF patients.

The purpose of this study is to determine the various factors that cause shortness of breath (or dyspnea) in patients with CF and to determine how treatment with Orkambi can manipulate these factors to improve shortness of breath and exercise capacity. The investigators hypothesize that lumacaftor/ivacaftor will reduce dyspnea intensity ratings and improve exercise capacity. These improvements will be associated with improvements in the ventilatory response to exercise.

Exercise capacity is an important outcome parameter in CF and is a strong predictor of disease prognosis including survival. While previous studies have reported improved respiratory symptoms in CF patients taking Orkambi, it remains uncertain as to whether this translates into improvements in exercise performance. Furthermore, the improvement in lung function parameters observed in these studies evaluating Orkambi in CF were modest compared to ivacaftor in CF and therefore stressing the respiratory system to its physiologic limits through exercise might provide a more sensitive outcome measure to evaluate the response to the Orkambi treatment option.

The objective of this study is to perform detailed cardiopulmonary exercise testing before and after the initiation of lumacaftor/ivacaftor to evaluate its effect on exertional dyspnea and exercise capacity, and to evaluate potential physiological mechanisms of improvement in patients with CF.

Experimental Overview: Participants with CF will report to the laboratory on four separate visits. Visit 1 and 2 will occur before the participants go on drug (Orkambi) and will be separated by a minimum of 2 days between visits. Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. On visit 1, participants will complete medical history screening, anthropometric measurements, pulmonary function assessment, and a symptom limited incremental cycle exercise test to determine peak incremental work rate. On visit 2, participants will complete chronic activity-related dyspnea, quality of life, and physical activity questionnaires, perform pulmonary function testing followed by a constant-load cycle exercise test at 80% of peak incremental work rate. Visits 3 and 4 will include chronic activity-related dyspnea, quality of life, and physical activity questionnaires, pulmonary function testing, and a constant-load cycle exercise test at 80% of peak incremental work rate. Detailed physiological and sensory measurements will be obtained during the exercise test sessions. Data from the constant-load cycle exercise tests performed on visits 2, 3, and 4 will address our hypothesis.

Exercise Protocol: All exercise testing will occur in the Cardiopulmonary Exercise Physiology Laboratory (CPEP lab). The CPEP lab is located on the 4th floor of the Burrard Building at St. Paul's Hospital (Vancouver, BC). A symptom-limited incremental exercise test will be performed on visit 1 using an electronically braked cycle ergometer (Ergoslect 200P; Ergoline GmbH, Bitz, Germany) according to recommended guidelines. The test will consist of steady-state rest for 6 minutes, a 1 minute warm-up of unloaded pedaling, and 15 watt stepwise increases in work rate every 2 minutes until symptom-limitation. Constant-load exercise tests on visits 2, 3, and 4 will include rest and warm-up periods followed by an immediate increase in work rate to 80% of maximal work (determined on visit 1) until symptom limitation.

Pulmonary Function: Spirometry, plethysmography, diffusing capacity of the lung for carbon monoxide (DLCO), maximum respiratory pressures, and impulse oscillometry will be performed on all study visits according to standard recommendations. A commercially available cardiopulmonary testing system will be used, and all measurements will be expressed as % of predicted normal values.

Dyspnea Evaluation: Dyspnea intensity (defined as "the sensation of laboured or difficult breathing") and perceived leg discomfort will be evaluated at rest, every minute during exercise, and at peak exercise using the modified 10-point Borg scale on all testing visits. Participants will be asked to describe their dyspnea during exercise after the intensity ratings at end-exercise using the following 3 descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all 3 of the descriptors can be chosen at any one time. Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire.

Cardio-respiratory Responses to Exercise: Standard cardio-respiratory measures will be recorded on a breath-by-breath basis and averaged over 30-second epochs, including minute ventilation (V'E), oxygen consumption (VO2), carbon dioxide production (CO2), tidal volume, and breathing frequency using a commercially available metabolic cart. Operating volumes (i.e., end-expiratory and end-inspiratory lung volumes) will be derived from dynamic inspiratory capacity (IC) manoeuvres as previously described. For safety purposes, electrocardiography will be monitored using a 12-lead electrocardiogram (ECG), blood pressure will be measured using a manual sphygmomanometer, and arterial oxygen saturation will be monitored using pulse oximetry. All exercise tests will be administered by experienced exercise physiologists. All exercise tests will be supervised by either Dr. Quon, Dr. Wilcox, Dr. Goodwin or another qualified physician. Exercise tests will be terminated based on established criteria as per American College of Sports Medicine guidelines.

Computed Tomography Phenotyping: Existing chest computed tomography (CT) scans, obtained through routine clinical practice, will be used for descriptive exploratory purposes to examine the relationship between the extent of bronchiectasis vs. mucus plugging vs. air trapping (based on CF-specific CT scoring) on the physiological and sensory responses to exercise in patients with CF.

Clinical Data Collection: The following clinical data (collected as part of routine clinical care) will be obtained via chart review: Medication review (Visit 1), Co-morbidities (Visit 1), Respiratory microbiology (Visit 1), Sweat Chloride (Visits 1, 3 and 4).

Study Participants: The study will include 16 participants in total. Participants satisfying inclusion and exclusion criteria will be recruited from the University of British Columbia Adult CF Clinic located on the 8th floor of the Providence Building within the Division of Respiratory Medicine at St. Paul's Hospital.

Statistical Analysis: Data will be presented as means ± standard deviation unless otherwise specified. Within-group comparison of exercise responses during constant-load exercise tests will be performed using paired t-tests with Bonferroni corrections where appropriate, comparing exercise responses during constant-load exercise tests performed before (visit 2) and after (visits 3 and 4) initiating full dose of Orkambi. Within-group comparison of exertional dyspnea will be based on Borg dyspnea ratings taken at iso-time, defined as the maximum time achieved on constant-load exercise tests performed on visits 2, 3, and 4. An additional analysis will include adjustment for potential covariates including age, sex, and baseline lung function (FVC and DLCO). Pearson correlation coefficients will be used to examine the association between measured variables (e.g. breathing patterns, ventilatory responses, operating lung volumes, pulmonary function variables, etc.) with changes in Borg ratings and endurance time. Reasons for stopping exercise and qualitative descriptors of dyspnea will be analyzed as frequency statistics and compared between constant -load exercise tests performed on visits 2, 3, and 4 using the McNemar's test at iso-time. A P-value less than 0.05 will be regarded as statistically significant. Statistical analysis of the data will be performed using Stata v11.2 (StataCorp, Texas, USA).

Sample Size and Power Calculation: A sample size of 16 per group provides 80% power to detect a 1 Borg unit difference between groups in dyspnea intensity at a standardized work rate during incremental cycle exercise, based on a standard deviation of 1 unit, α=0.05 and a 2-tailed test of significance. This sample size is also adequate to detect statistically significant differences in our other outcomes (operating lung volumes) based on previous studies in humans.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF and homozygous for the F508del mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
* Plan to initiate Orkambi™ by the treating physician within 30 days of the enrolment visit
* Aged 19 years or older
* Stable clinical status based on clinical judgment of the treating physicians (Drs Wilcox, Quon or Goodwin)
* Forced Expiratory Volume in 1 second (FEV1.0) < 90% predicted
* Body mass index greater than 16 or less than 30 kg/m2
* Currently non-smoking or a past smoking history of less than 20 pack-years
* Able to read and understand English

Exclusion Criteria:

* A disease other than CF that could importantly contribute to dyspnea or exercise limitation
* Chronic airway infection with Mycobacterium abscessus, Burkholderia cepacia complex, or other organisms with infection control implications based on the treating physicians
* Contraindications to clinical exercise testing
* Use of supplemental oxygen or desaturation less than 85% with exercise
* Diagnosis of pneumothorax in the past 4 weeks
* History of organ transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CF patients will be recruited from the St. Paul's Hospital UBC Adult CF Clinic.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-07; Primary Completion 2019-12 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in iso-time dyspnea rating from baseline (visit 2) to visit 3 and 4 during constant-load exercise tests. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Dyspnea rating measured using the Borg 0-10 category ratio scale.

SECONDARY OUTCOMES:
Change from baseline cardio-respiratory responses during constant-load exercise tests (prior to Orkambi initiation to full dose) at 1 and 3 months after initiating full dose of Orkambi. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Cardio-respiratory responses include exercise endurance time, minute ventilation, oxygen consumption, carbon dioxide production, ventilatory equivalents for oxygen and carbon dioxide, tidal volume, breathing frequency, and operating lung volumes.
Change from baseline chronic activity-related dyspnea (prior to Orkambi initiation to full dose) at 1 and 3 months after initiating full dose of Orkambi. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Chronic activity-related dyspnea measured using the Modified Baseline Dyspnea Index, Baseline and Transition Dyspnea Index, Modified Medical Research Council Dyspnea Scale, and Oxygen Cost Diagram.
Change from baseline quality of life (prior to Orkambi initiation to full dose) at 1 and 3 months after initiating full dose of Orkambi. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Quality of life measured using the St. George's Respiratory Questionnaire.
Change from baseline physical activity (prior to Orkambi initiation to full dose) at 1 and 3 months after initiating full dose of Orkambi. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Physical activity measured using the International Physical Activity Questionnaire (long version) and Recent Physical Activity Questionnaire.
Change from baseline pulmonary function measures (prior to Orkambi initiation to full dose) at 1 and 3 months after initiating full dose of Orkambi. | Parameters will be measured during 3 visits. Visit 2 will occur before the participants go on drug (Orkambi). Visit 3 and 4 will occur at 1 month and 3 months after initiating full dose of drug, respectively. All visits will be completed within 4 months.
  Pulmonary function measures include spirometry, plethysmography, diffusing capacity of the lung for carbon monoxide, maximum respiratory pressures, and impulse oscillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia - Centre for Heart Lung Innovation
Locations (1):
- UBC James Hogg Research Centre, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Quon BS, Ramsook AH, Dhillon SS, Mitchell RA, Boyle KG, Wilcox PG, Guenette JA. Short-term effects of Lumacaftor/Ivacaftor (Orkambi) on exertional symptoms, exercise performance, and ventilatory responses in adults with cystic fibrosis. Respir Res. 2020 Jun 1;21(1):135. doi: 10.1186/s12931-020-01406-z. PMID 32487229